CLINICAL TRIAL: NCT06444776
Title: Therapy-Associated Saliva and Taste Change Evaluation (TASTE) in Head & Neck Cancer
Brief Title: Therapy-Associated Saliva and Taste Change Evaluation (TASTE) in Head & Neck Cancer Patients Undergoing Radiotherapy
Acronym: TASTE
Status: Recruiting | Type: Observational
Sponsor: Sonja Stieb, MD (Other)
Collaborators: Kantonsspital Aarau (Other); University of Bern (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Sonja Stieb, MD, Dr. med. Sonja Stieb, MD, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Other Study IDs: 2022-00706
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy; Taste impairment; Dysgeusia; Xerostomia; Saliva; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Dysgeusia; Xerostomia | interventions — Smell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer patients referred for radiation therapy
  Interventions: Diagnostic Test: Repetitive (semi-)objective and subjective taste, smell, and saliva analysis

INTERVENTIONS:
Diagnostic Test: Repetitive (semi-)objective and subjective taste, smell, and saliva analysis — Study participants will undergo repetitive assessments of their taste, smell and saliva, using quality of life questionnaires, taste strips, sniffin sticks, and analysis of salivary function and composition.
  Assessments will be done before treatment, in the 4th week (+/- 1 week) and last week of radiation therapy (+/- 1 week), and at 6 months (+/- 1 months) and 1 and 2 years post-therapy (+/- 3 months).
  At the minimum, participants are expected to complete the assessments at baseline and 1 year after the end of radiation therapy. Assessments at all other time points are strongly encouraged but will be optional.

SUMMARY:
One of the main side effects of radiation therapy to the head and neck region is altered taste sensation. This causes significant morbidity and has profound effects on the quality of life (QoL) of patients. While radiation-associated toxicities like xerostomia and dysphagia are part of large investigations, data on taste impairment is sparse.

The TASTE study sets out to further our understanding of this common side effect with the goal to prevent radiation-associated taste impairment in future patients.

In this prospective, observational multicenter study 150 head and neck cancer patients undergoing radiation therapy will be recruited. Participants will undergo repetitive (semi-) objective and subjective assessment of their taste, smell and salivary function at specific time points before, during and after radiotherapy. Primary endpoint will be patient-reported taste impairment 12 months post radiation therapy using a standardized quality of life questionnaire (MDASI-HN). Secondary endpoints will include taste impairment measured using taste strips at 12 months and 2 years post radiation therapy. Differences between subgroups (radiation side, chemotherapy, etc.) and changes over time will be assessed while adjusting for confounding factors (e.g. age, sex, smoking history). Based on the aquired data, a normal tissue complication probability model for late radiation-associated taste impairment will be develeoped.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients
* Referred for radiation therapy with curative intent, both definitive and post-operative
* Age ≥18
* Karnofsky performance index of at least 50%
* Anticipated mean radiation dose to the taste bud bearing tongue mucosa or at least one of the major salivary glands (parotid, submandibular, and/or sublingual gland) of at the minimum 5 Gy

Exclusion Criteria:

* Pregnancy
* Pre-existing subjective complete loss of taste before start of radiation therapy
* Planning CT and radiation therapy with oral stent or spacer
* Partial or total glossectomy which impairs taste assessments of at least one side of the tongue or impairs contouring of the taste bud bearing tongue mucosa on the planning CT
* Inability to follow instructions related to study procedures or inability to fill in the questionnaires
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult head and neck cancer patients referred for radiation therapy with curative intent, both definitive and post-operative
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Taste impairment | 12 months post-treatment
  Patient-reported taste impairment assessed by the MDASI-HN (MD Anderson Symptom Inventory Head and Neck module) questionnaire

SECONDARY OUTCOMES:
Taste impairment | 24 months post-treatment
  Patient-reported taste impairment assessed by the MDASI-HN (MD Anderson Symptom Inventory Head and Neck module) questionnaire
Taste impairment | 12 and 24 months post-treatment
  Taste impairment diagnosed using taste strips

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Kantonsspital Aarau, Zentrum für Radio-Onkologie KSA-KSB, Aarau, Canton of Aargau
  - Universitätsspital Bern, Bern
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No